CLINICAL TRIAL: NCT06885411
Title: Ototixicity in Patients With a Metal-on-Metal Hip Arthroplasty
Brief Title: Ototoxicity in Patients With MoM Hip Bearings
Acronym: GODMOTHER
Status: Recruiting | Type: Observational
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Collaborators: Reinier de Graaf Groep (Other); Erasmus Medical Center (Other); Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: OC-2021-012
Record Dates: First submitted 2024-11-20; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Ototoxic Hearing Loss; Cobalt Poisoning; Chromium Causing Toxic Effect; Arthroplasty Complications
Keywords: Metal-on-Metal implant; Cobalt; Chromium; Hip arthroplasty; auditory system; Otoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Bloodsample to determine cobalt and chromium concentrations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Arthroplasty patients: Patients with a (revised) metal-on-metal hip arthroplasty
  Interventions: Other: metal-on-metal hip arthroplasty

INTERVENTIONS:
Other: metal-on-metal hip arthroplasty — Cobalt and chromium release from metal-on-metal hip arthroplasties.

SUMMARY:
The goal of this observational study is to learn about ototoxicity in patients with a MoM hip arthroplasty. The main question it aims to answer is:

• What is the prevalence of hearing loss in patients with high and low plasma metal concentrations.

ELIGIBILITY:
Inclusion Criteria:

* all MoM patients from the different clinics
* revision MoM
* willing to participate
* speak/write the Dutch language

Exclusion Criteria:

* Not willing to participate
* previous ENT surgery or ENT pathology

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients in the participating hospitals with a MoM hip arthroplasty or a revised MoM hip arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Mid frequency hearing loss | Participants will perform a hearing test once during the study, during a visit of the outpatient clinic.
  Mid frequency hearing loss will be determined once with a conventional pure-tone audiometry test during a visit of the outpatient clinic

SECONDARY OUTCOMES:
Age | Age will be determined once for each participant, at time of the visit of the outpatient clinic
  Age will be determined once, during a visit of the outpatient clinic
subjective general health and subjective hearing loss measured with the Amsterdam Inventory for Auditory Disability and Handicap questionnaire. | The questionnaire will be completed once by each participant, at time of the visit of the outpatient clinic
  The subjective general health and subjective hearing loss will be determined by Amsterdam Inventory for Auditory Disability and Handicap. The questionnaire will be completed by the participants once,at time of the visit of the outpatient clinic
BMI | Lenght and weight will be determined once for each participant, at time of the visit of the outpatient clinic
  BMI will be dermined once, at time of measurement weight and height will be combined to report BMI in kg/m^2
Cobalt serum concentration | Cobalt serum concentration will be determined once for each participant, at time of the visit of the outpatient clinic
  Cobalt serum concentration will be dermined once, throught venipuncture, at time of the visit of the outpatient clinic.
Chromium serum concentration | Chromium serum concentration will be determined once for each participant, at time of the visit of the outpatient clinic
  Chromium serum concentration will be dermined once, throught venipuncture, at time of the visit of the outpatient clinic.

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier de Graaf Ziekenhuis, Delft, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT06885411/Prot_SAP_000.pdf